CLINICAL TRIAL: NCT03116191
Title: Trial of SK-1404 for Nocturia Due to Nocturnal Polyuria in Japanese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VA1001
Record Dates: First submitted 2017-04-06; First posted 2017-04-14 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Nocturia Due to Nocturnal Polyuria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SK-1404 high dose (Experimental)
  Interventions: Drug: SK-1404
- SK-1404 middle dose (Experimental)
  Interventions: Drug: SK-1404
- SK-1404 low dose (Experimental)
  Interventions: Drug: SK-1404
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SK-1404 — 4 weeks of repeated administration of SK-1404 to the patients of nocturia
  Arms: SK-1404 high dose; SK-1404 low dose; SK-1404 middle dose
Drug: Placebo — 4 weeks of repeated administration of Placebo to the patients of nocturia
  Arms: Placebo

SUMMARY:
The purpose of this trial is to demonstrate efficacy of SK-1404 against placebo for the treatment of subjects with nocturia due to nocturnal polyuria, during 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 5 > nocturnal voids ≥2
* NPI >0.33

Exclusion Criteria:

* Polydipsia
* Cardiac failure
* Syndrome of inappropriate antidiuretic hormone secretion
* Hyponatraemia
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Moderate or severe over-active bladder (OAB)
* Severe benign prostate hyperplasia (BPH)
* Sleep apnoea
* Interstitial cystitis
* Stress urinary incontinence
* Diabetes insipidus
* Complication or a history of urological cancer

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of nocturnal voids | 4 weeks
  Assessed by the voiding diary

SECONDARY OUTCOMES:
Change from base line in mean nocturnal urine volume | 4 weeks
  Assessed by the voiding diary
Change from base line in mean time to first awakening to void | 4 weeks
  Assessed by the voiding diary
Change from base line in mean Nocturnal Polyuria Index (NPI) | 4 weeks
  Assessed by the voiding diary
Change from base line in the score of Nocturia-Specific Quality-of-Life Questionnaire (N-QoL) | 4 weeks
  Assessed by the voiding diary

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan